CLINICAL TRIAL: NCT04023214
Title: Endothelial Dysfunction in Autosomal Dominant Polycystic Kidney Disease
Brief Title: The Role of Endothelial Dysfunction in Adult Polycystic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH15983
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Polycystic Kidney, Autosomal Dominant
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- ADPKD: ADPKD patients
  Interventions: Diagnostic Test: Peripheral (digital) arterial tonometry
- Controls: Healthy volunteers
  Interventions: Diagnostic Test: Peripheral (digital) arterial tonometry

INTERVENTIONS:
Diagnostic Test: Peripheral (digital) arterial tonometry — This will be measured using the EndoPAT system (Itamar Medical)

SUMMARY:
This pilot study will compare endothelial function in patients with ADPKD with matched healthy volunteers and normotensive chronic kidney disease stage 1 & 2 patients. Patients will undergo a single assessment of endothelial function and measurement of plasma and urine levels of biomarkers of endothelial function.

DETAILED DESCRIPTION:
Following recruitment we will record the following baseline demographics; age, gender, smoking status, body mass index, medical history.

Participants will undergo a noninvasive vascular assessment, venepuncture and will provide a urine sample.This will be done during a single visit to the CRF.

Noninvasive vascular assessment will consist of:

1. Peripheral Arterial Tonometry This will be measured using the EndoPAT system (Itamar Medical)

   Endothelial shear stress flow stimulus will be provided by inflation of a blood pressure cuff around the upper non-dominant arm to suprasystolic pressure (but <300mmHg) for 5 minutes. Following release of the cuff the resulting digital microcirculation vasodilatory response to ischaemic hyperaemia, quantified as the pulse wave amplitude, will be monitored over 5 minutes. The peak pulse wave amplitude measured at 90-150s post cuff deflation relative to baseline will be indexed to the changes in the opposite arm to give the reactive hyperaemia index. This measure of endothelial function constitutes the outcome measure.
2. Blood Pressure Assessment Brachial artery blood pressure will be measured in the left arm in the supine position using an automated device (Dinamap) and in accordance with the clinical research facility SOP.
3. Blood samples and urine samples

Samples for plasma will be centrifuged and stored at -80C. Biochemical analysis will be performed by the laboratory of the STH NHS Trust for standard tests and by validated assays for non-routine markers (as detailed below) in the Academic Nephrology Unit.

Participants will be asked to collect a 24h urine sample from the day before the study visit and to provide a spot urine sample on the day. This will be analysed at the laboratory of the STH NHS Trust.

Biochemical Analysis

Serum samples will be analyzed for Full blood count, Urea, Electrolytes, Glucose, Insulin, Lipid Profile, Homocysteine, (Hs) CRP and Creatinine Levels.

Serum and plasma will also be stored for future analysis of relevant biomarkers of endothelial function or nitric oxide metabolism as indicated by preliminary results.

Urine samples will be analysed initially for protein creatinine ratio (PCR). The rest will be frozen for future analysis of urinary biomarkers of endothelial function or nitric oxide metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Age >18yrs, <50yrs
* Able to understand spoken/written English sufficiently to give informed consent and to take part in clinical assessment
* Clinical diagnosis of ADPKD
* eGFR >60ml/min/1.73m2

Exclusion Criteria:

* No history of cardiovascular disease or hypertension
* Not diabetic
* Not smoking
* Not breastfeeding
* Not pregnant
* Not taking any regular medication (except oral contraceptives)
* No musculoskeletal conditions contraindicating inflation of a blood pressure cuff to suprasystolic pressures around the forearm (as part of EndoPAT measurements)
* Not morbidly obese: BMI<35 (May contribute to endothelial dysfunction)
* eGFR <60ml/min/1.73m2

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normotensive ADPKD patients with well preserved GFR (>60ml/min) ie those with Stage 1 or 2 Chronic Kidney Disease recruited from a specialist PKD clinic. Healthy controls will be recruited matched to age, sex, body mass index (BMI) and eGFR of the ADPKD patients.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-07-25 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Reactive hyperemia index (RHI) | Baseline
  EndoPAT values (Endoscore)

SECONDARY OUTCOMES:
Systolic and diastolic Blood pressure | Baseline
  mm Hg
Proteinuria | Baseline
  Protein creatinine ratio

CONTACTS AND LOCATIONS:
Overall Officials: Albert Ong, Principal Investigator — STH; Timothy Chico, Study Director — STH

IPD SHARING:
Plan to Share IPD: No